CLINICAL TRIAL: NCT02797977
Title: A Phase 1/2 Trial of Oral SRA737 (a Chk1 Inhibitor) Given in Combination With Gemcitabine Plus Cisplatin or Gemcitabine Alone in Subjects With Advanced Cancer
Brief Title: A Phase 1/2 Trial SRA737 in Combination With Gemcitabine and Cisplatin or Gemcitabine Alone in Advanced Cancer Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sierra Oncology LLC - a GSK company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SRA737-02
Record Dates: First submitted 2016-05-23; First posted 2016-06-14 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2022-06

CONDITIONS: Advanced Solid Tumors
Keywords: Replication Stress; Advanced solid tumors; CCNE1; TP53; BRCA1; BRCA2; MYC; RAD50; Fanconi anemia; Cell Cycle; High grade serious ovarian cancer; Small cell lung cancer; Soft tissue sarcoma; Cervical/anogenital cancer; Phase 1; Phase 2; Dose escalation; Chk1 inhibitor; Checkpoint Kinase 1; Synthetic lethality; Next-Generation Sequencing; Genetic biomarkers
MeSH Terms: conditions — Fanconi Anemia; Small Cell Lung Carcinoma; Sarcoma | interventions — SRA737; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard-Dose Triplet Combination (Experimental): SRA737 will be administered orally on Days 2, 3, 9, and 10 of each 21-day cycle. Subjects will receive a single dose of SRA737 between 4 to 7 days prior to starting the first cycle for PK profiling. Gemcitabine will be administered intravenously on Days 1 and 8 of each 21-day cycle. Cisplatin will be administered on Day 1 of each 21-day cycle. Subjects can continue taking the study treatment if they are safely receiving clinical benefit and able to follow the requirements of the study.
  Interventions: Drug: SRA737, gemcitabine, cisplatin
- Low-Dose Gemcitabine Combination (Experimental): SRA737 will be administered orally on Days 2, 3, 9, 10, 16, and 17 of each 28-day cycle. Subjects will receive a single dose of SRA737 between 4 to 7 days prior to starting the first cycle. Gemcitabine will be administered intravenously on Days 1, 8, and 15 of each 28-day cycle. Subjects can continue taking the study treatment if they are safely receiving clinical benefit and able to follow the requirements of the study.
  Interventions: Drug: SRA737, gemcitabine

INTERVENTIONS:
Drug: SRA737, gemcitabine, cisplatin
  Arms: Standard-Dose Triplet Combination
Drug: SRA737, gemcitabine
  Arms: Low-Dose Gemcitabine Combination

SUMMARY:
The purpose of this clinical study is to establish the safety profile, determine the maximum tolerated dose (MTD) and recommend a Phase 2 dose (RP2D) and schedule of SRA737 in combination with low dose gemcitabine; and to evaluate the efficacy of SRA737 in combination with low dose gemcitabine in prospectively-selected subjects with genetically-defined tumors that have predicted sensitivity to Chk1 inhibition based on factors including: genetic profiling of tumor tissue or ctDNA, HPV status, and germline BRCA1 and BRCA2 gene status. Specific cancer indications that frequently feature these factors will be studied.

Preclinical and clinical data support the hypothesis that active doses of SRA737 may be strongly potentiated by sub-therapeutic doses of gemcitabine, which should lead to clinical efficacy. To test this hypothesis, SRA737 in combination with low dose gemcitabine is being explored in this study.

DETAILED DESCRIPTION:
SRA737 is a potent, highly selective, orally bioavailable small molecule inhibitor of Chk1, a key regulator of cell cycle progression and the DNA Damage Response (DDR) replication stress response. In cancer cells, intrinsic replication stress (RS) is induced by factors such as oncogenes (e.g., CCNE1 or MYC), genetic mutations in DNA repair machinery (e.g., BRCA1 or FA), genetic mutations leading to a dysregulated cell cycle (e.g., TP53 or RAD50) or other genomic alterations. This replication stress results in persistent DNA damage and genomic instability leading to an increased dependency on Chk1 for survival. Targeted inhibition of Chk1 by SRA737 may therefore be synthetically lethal to cancer cells with elevated intrinsic RS.

The critical role of Chk1 in mediating cellular responses to RS affords the opportunity to combine SRA737 with sub-therapeutic concentrations of the RS-inducing agent gemcitabine. Low concentrations of gemcitabine cause a prolonged cell cycle S-phase and induce hallmarks of RS without inducing overt cytotoxicity. Gemcitabine profoundly depletes DNA replication building blocks and targets proliferating cells by inducing RS through induction of stalled replication forks. In response, Chk1 has an important role in stabilizing and preserving replication fork complexes in the context of RS, preventing catastrophic replication fork collapse and double strand breaks. Extensive preclinical data, as well as clinical data, support the synergistic interaction between Chk1 inhibition and gemcitabine.

The purpose of this clinical study is to: establish the safety profile, determine the MTD, and propose a RP2D and schedule for SRA737 in combination with low dose gemcitabine. In addition, the study aims to evaluate the preliminary efficacy of SRA737 in combination with low dose gemcitabine in prospectively-selected subjects with tumors that have predicted sensitivity to Chk1 inhibition.

This clinical study consists of three phases:

1. A Standard-Dose Triplet Combo Dose Escalation Phase 1. This phase, which has concluded, evaluated a triplet combination of SRA737 with standard-dose gemcitabine and cisplatin in subjects with solid tumors.
2. A Low-Dose Gemcitabine Combo Dose Escalation Phase 1. Cohorts of 3 to 6 subjects are being given escalating doses of SRA737 on an intermittent schedule in addition to low dose gemcitabine until the combination MTD is reached. The dose or frequency of gemcitabine may also be reduced during this process and alternative dosing schedules for SRA737 may be considered. When the MTD or a minimum efficacious dose range has been achieved for SRA737, or when evidence of anti-tumor activity is observed, the gemcitabine dose may be escalated with corresponding decreases in the SRA737 dose as necessary for safety.
3. A Low-Dose Gemcitabine Combo Cohort Expansion Phase 2. After the MTD and/or RP2D has been identified, the trial will explore the preliminary efficacy of SRA737 plus low dose gemcitabine in prospectively-selected subjects with tumors that harbor genomic alterations linked to increased replication stress and that are hypothesized to be more sensitive to Chk1 inhibition via synthetic lethality. Enrollment for expansion cohorts may alternatively begin prior to the completion of dose escalation and determination of MTD or RP2D, if there is evidence of anti-tumor activity or if the minimal plasma concentration of SRA737 is maintained above a threshold at which sustained Chk1 inhibition is anticipated at 24 hours after dosing.

This phase is targeting enrollment of genetically-selected patients into four expansion cohorts from specific indications that are predicted to have a high prevalence of such alterations, including locally advanced or metastatic:

* high-grade serous ovarian cancer (HGSOC),
* small cell lung cancer (SCLC);
* soft tissue sarcoma (STS); and
* cervical/anogenital cancer.

To qualify for enrolment into these cohorts, the subject's tumor must have evidence of predicted sensitivity to Chk1 inhibition based on factors including:

* For subjects with HGSOC, documented somatic or germline BRCA1 and BRCA2 wild-type status will confer eligibility without requirement for prospective genetic profiling. If documented BRCA status is not available, genetic profiling may be performed prospectively to determine eligibility.
* Subjects with SCLC are eligible without requirement for prospective genetic profiling on the basis of very high prevalence of cancer related alterations in the tumor suppressor genes (eg, TP53 and RB1) in this population.
* For subjects with STS, and any others for whom genetic profiling is performed prospectively, eligibility will be determined by the sponsor's review of genetic abnormalities detected in genes in the following categories:

  * Key tumor suppressor genes regulating G1 cell cycle progression/arrest such as RB1, TP53, etc.
  * The DNA damage response pathway including ATM, BRCA1, BRCA2, mismatch repair genetic alterations and/or high microsatellite instability.
  * Genetic indicators of replicative stress such as gain of function/amplification of Chk1 or ATR or other related gene.
  * Oncogenic drivers such as MYC, CCNE1, etc.
* For subjects with anogenital cancer, known HPV positive status will confer eligibility without requirement for prospective genetic profiling. If HPV status is not known or not positive, genetic profiling (or HPV testing where appropriate) may be performed prospectively to determine eligibility. Subjects with cervical cancer or squamous cell carcinoma of the anus are eligible without requirement for prospective genetic profiling based on the very high prevalence of HPV positivity in these populations.

Tumor genetics will be determine using Next-Generation Sequencing.

ELIGIBILITY:
Key Inclusion Criteria:

1. For Dose Escalation: subjects with locally advanced or metastatic, histologically or cytologically proven solid tumor, relapsed after or progressing despite conventional treatment
2. Life expectancy of at least 12 weeks
3. World Health Organization (WHO) performance status of 0-1
4. Must meet select hematological and biochemical laboratory indices
5. Archival tumor tissue or accessible tumor and willingness to consent to a biopsy

Expansion Only:

1. Histologically or cytologically proven advanced malignancy of the following types, for which no other conventional therapy is considered appropriate:

   * High-grade serous ovarian cancer (HGSOC)
   * Small cell lung cancer
   * Soft tissue sarcoma
   * Cervical/anogenital cancer
2. Measurable disease per RECIST v1.1
3. Subjects must have predicted sensitivity to Chk1 inhibition based on factors including: genetic profiling of tumor tissue or ctDNA, HPV status, and germline BRCA1 and BRCA2 gene status. All subjects will have genetic profiling from tumor tissue or ctDNA; profiling will be performed prospectively if required to evaluate Chk1 sensitivity or otherwise performed retrospectively.

   1. For subjects with HGSOC, documented somatic or germline BRCA1 and BRCA2 wild-type status will confer eligibility without requirement for prospective genetic profiling. If documented BRCA status is not available, genetic profiling may be performed prospectively to determine eligibility.
   2. Subjects with SCLC are eligible without requirement for prospective genetic profiling on the basis of very high prevalence of cancer related alterations in the tumor suppressor genes (eg, TP53 and RB1) in this population.
   3. For subjects with STS, and any others for whom genetic profiling is performed prospectively, eligibility will be determined by the sponsor's review of genetic abnormalities detected in genes in the following categories:

      Key tumor suppressor genes regulating G1 cell cycle progression/arrest such as RB1, TP53, etc. For relevant cancers, positive human papilloma virus (HPV) status is also considered for eligibility.
      * The DNA damage response pathway including ATM, BRCA1, BRCA2, mismatch repair genetic alterations and/or high microsatellite instability.
      * Genetic indicators of replicative stress such as gain of function/amplification of Chk1 or ATR or other related gene.
      * Oncogenic drivers such as MYC, CCNE1, etc.
   4. For subjects with anogenital cancer, known HPV positive status will confer eligibility without requirement for prospective genetic profiling. If HPV status is not known or not positive, genetic profiling (or HPV testing where appropriate) may be performed prospectively to determine eligibility. Subjects with cervical cancer or squamous cell carcinoma of the anus are eligible without requirement for prospective genetic profiling based on the very high prevalence of HPV positivity in these populations.

Key Exclusion Criteria:

1. Received the following prior or current anticancer therapy in the timeframes noted prior to receiving SRA737 and have recovered from toxicity:

   1. Radiotherapy, chemotherapy, PARP inhibitors, other targeted therapies, or other IMPs within 2 weeks
   2. Nitrosoureas or Mitomycin C within 6 weeks
   3. Any prior treatment with a Chk1 inhibitor at any point or prior treatment with an ATR inhibitor within 6 months
2. No more than 3 previous treatment regimens for advanced disease (not applicable to HGSOC expansion cohort)
3. Other malignancy within the past 2 years, except for adequately treated tumors
4. If, in the opinion of the Investigator, the subject is highly likely to experience clinically significant myelosuppression
5. Ongoing toxic manifestations of previous treatments greater than NCI-CTCAE Grade 1
6. History of allergy to gemcitabine
7. New or progressing brain metastases. Subjects with brain metastases that have been asymptomatic and radiologically stable over an 8-week period and have not been treated with steroids during that time may be included with approval from the sponsor.
8. High medical risk because of nonmalignant systemic disease
9. Serologically positive for hepatitis B, hepatitis C or HIV
10. Serious cardiac condition, left ventricular ejection fraction < 45% at baseline, history of cardiac ischemia within the past 6 months, or prior history of cardiac arrhythmia requiring treatment, unless approved by the sponsor.
11. Prior bone marrow transplant or extensive radiotherapy to greater than 25% of bone marrow within the previous 8 weeks
12. Peanut allergy
13. QTcF > 450 msec in adult makes and > 470 msec in adult females
14. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of SRA737
15. Inability to swallow capsules without chewing or crushing
16. Is a participant or plans to participate in another interventional clinical trial
17. Any other condition which in the Investigator's opinion would not make the subject a good candidate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-04-08 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events as assessed by CTCAE4.03 | Up to 30 days after last dose of SRA737
Maximum tolerated dose of SRA737 administered in combination with gemcitabine | Cycle 1 (28 days) in the Dose Escalation Phase
Recommended Phase 2 dose of SRA737 in combination with gemcitabine. | Up to 30 days after last dose of SRA737

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Sierra Oncology LLC - a GSK company
Locations (20):
- Spain (6):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - START Madrid, Madrid
  - Hospital Universitario 12 de Octobre, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Biomedical Research Institute INCLIVA, Valencia
- United Kingdom (14):
  - Royal Marsden Hospital, Sutton, London
  - Belfast City Hospital, Belfast, Northern Ireland
  - Oxford University Hospitals, Headington, Oxford
  - Velindre Cancer Centre, Cardiff, Whitchurch
  - The Clatterbridge Cancer Centre, Bebington, Wirral
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - Leeds Teaching Hospital of St James University Hospital, Leeds
  - University Hospital of Leceister NHS TRUST, Leicester
  - Guy's and St Thomas', London
  - Sarah Cannon Research Institute, London
  - University College London, London
  - The Christie NHS Foundation Trust, Manchester
  - Freeman Hospital, Newcastle upon Tyne
  - Sheffield Teaching Hospitals, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jones R, Plummer R, Moreno V, Carter L, Roda D, Garralda E, Kristeleit R, Sarker D, Arkenau T, Roxburgh P, Walter HS, Blagden S, Anthoney A, Klencke BJ, Kowalski MM, Banerji U. A Phase I/II Trial of Oral SRA737 (a Chk1 Inhibitor) Given in Combination with Low-Dose Gemcitabine in Patients with Advanced Cancer. Clin Cancer Res. 2023 Jan 17;29(2):331-340. doi: 10.1158/1078-0432.CCR-22-2074. PMID 36378548

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-03): https://cdn.clinicaltrials.gov/large-docs/77/NCT02797977/Prot_SAP_000.pdf